CLINICAL TRIAL: NCT00574184
Title: Pelvic Angiography in Non-Responders to Phosphodiesterase-5 Inhibitors (PANPI)
Acronym: PANPI
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 200513528
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2008-03

CONDITIONS: Erectile Dysfunction
Keywords: ED; Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The specific aim of this pilot study is to describe the angiographic prevalence and pattern of internal pudendal artery (and associated inflow vessel) atherosclerosis in patients with erectile dysfunction who are non-responsive to PDE-5 inhibitors (i.e., Viagra) who are referred for clinically-indicated cardiac catheterization.

DETAILED DESCRIPTION:
The specific aim of this study is to determine if the deep penile arteries can be seen angiographically from the iliac arteries to delineate penile vasculature. Significant obstructive atherosclerotic disease of the deep penile arteries may be present in impotent males. The etiology of erectile dysfunction is multifactorial and may involve vascular disease, endocrine disorders, neurologic disease, prescription medications, psychological issues and/or trauma in any given patient. Vascular disease in patients with erectile dysfunction may be due to trauma, congenital anomalies, or atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* at least 50 years
* erectile dysfunction
* dissatisfaction with their use of a phosphodiesterase-5 inhibitor
* coronary artery disease (or at risk for coronary artery disease)
* undergoing diagnostic cardiac catheterization or patients with peripheral vascular disease undergoing peripheral arteriography

Exclusion Criteria:

* Patients who respond favorably to phosphodiesterase-5 inhibitors
* known non-vascular etiologies of their erectile dysfunction
* probable neurogenic erectile dysfunction due to radiation injury, surgery, or transurethral resection of the prostate
* calculated GFR < 60 ml/min/1.73 m2 will also be excluded
* disease that necessitates complex percutaneous intervention will be excluded per the investigators discretion

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will include males who are scheduled to undergo cardiac catheterization or peripheral arteriography at UC Davis Medical Center who have erectile dysfunction and poor response to oral phosphodiesterase-5 inhibitors (Viagra, Cialis and Levitra) as determined by their response to a standardized questionnaire. Dissatisfaction will be defined as a score of 21 or less on the ILEF-5 (International Index of Erectile Function questionnaire).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2005-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Distal aortography with iliofemoral run-off will be performed to evaluate disease in the common and internal iliac arteries. | During Procedural Cath

SECONDARY OUTCOMES:
Selective angiography of the internal pudendal artery (and accessory pudendal artery if present) will be performed bilaterally. | During Procedural Cath
Intra-arterial nitroglycerin (or papaverine or tolazoline if nitroglycerin is contraindicated) will be used to facilitate angiographic visualization of the internal pudendal and penile arteries. | During Procedural Cath

CONTACTS AND LOCATIONS:
Overall Officials: Jason Rogers, MD, Principal Investigator — University of California, Davis

REFERENCES:
- See also: UC Davis Health System — http://www.ucdmc.ucdavis.edu/clinicaltrials